CLINICAL TRIAL: NCT03018119
Title: Implementation of the National Partnership for Maternal Safety Obstetric Hemorrhage Bundle at a Tertiary Center: Utilization of the Delphi Method
Brief Title: Implementation of the NPMS Obstetric Hemorrhage Bundle at a Tertiary Center: Utilization of the Delphi Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Annemaria De Tina, Clinical Fellow - Obstetric Anesthesia, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015P002403
Record Dates: First submitted 2017-01-03; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Pregnancy Hemorrhage; Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Anesthesiologists (Active Comparator): Total: 11 Intervention: Survey
  Interventions: Other: Survey
- Obstetricians (Active Comparator): Total: 11 Intervention: Survey
  Interventions: Other: Survey
- Registered Nurses (Active Comparator): Total: 10 Intervention: Survey
  Interventions: Other: Survey
- Surgical Technicians (Active Comparator): Total: 6 Intervention: Survey
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey

SUMMARY:
The National Partnership for Maternal Safety (NPMS) developed an obstetric hemorrhage consensus bundle to provide every United States birthing facility consistent, validated practice guidelines. To facilitate implementation of each element of this bundle at the participants large tertiary center, the investigators utilized the Delphi method to identify deficiencies, perceived barriers to implementation, and multidisciplinary consensus on changes with high feasibility and impact on patient care.

ELIGIBILITY:
Inclusion Criteria:

* ≥ five years of experience on the L&D unit
* current employment on the L&D unit > 20h per week
* prior involvement in clinical obstetric hemorrhage situations

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Questionnaire of Obstetric Hemorrhage Bundle Components not Currently Adequately Implemented | 4 weeks

SECONDARY OUTCOMES:
Questionnaire of Perceived Barriers to Implementation of Obstetric Hemorrhage Bundle Components | 4 weeks
Questionnaire of Feasibility of Implementation of Obstetric Hemorrhage Bundle Components | 6 months
Questionnaire on Impact of Implementation of Obstetric Hemorrhage Bundle Components on Patient Care | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Farber, MD, MS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Main EK, Goffman D, Scavone BM, Low LK, Bingham D, Fontaine PL, Gorlin JB, Lagrew DC, Levy BS. National Partnership for Maternal Safety: consensus bundle on obstetric hemorrhage. Anesth Analg. 2015 Jul;121(1):142-148. doi: 10.1097/AOG.0000000000000869. PMID 26091046